CLINICAL TRIAL: NCT01184079
Title: Randomized Trial of Alternative HPV Vaccination Schedules in Males in a University Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Richard Zimmerman, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IISP#38206; PRO10070407 (Other: University of Pittsburgh IRB); I#0021806 (Other: University of Pittsburgh InfoEd)
Record Dates: First submitted 2010-08-11; First posted 2010-08-18 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Quadrivalent HPV Vaccine; Human Papillomavirus Vaccine
Keywords: human papillomavirus vaccine L1, type 6,11,16,18; HPV Vaccines; HPV L1 vaccine, quadrivalent 6,11,16,18
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12 months (Experimental): Administration of 3rd dose at 12 months quadrivalent human papillomavirus vaccine
  Interventions: Biological: quadrivalent human papillomavirus vaccine
- 6 month (Active Comparator): Administration of 3rd dose at 6 months quadrivalent human papillomavirus vaccine
  Interventions: Biological: quadrivalent human papillomavirus vaccine

INTERVENTIONS:
Biological: quadrivalent human papillomavirus vaccine — 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 12 months
  Other Names: Gardasil
  Arms: 12 months
Biological: quadrivalent human papillomavirus vaccine — 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 6 months
  Other Names: Gardasil
  Arms: 6 month

SUMMARY:
The investigators propose a randomized, open label trial of the immunogenicity of HPV vaccine among males 18-24 years old, comparing an on-time administration of the third dose with delayed administration of the third dose. All participants would receive the first and second doses according to schedule. They would be randomized to either Dose 3 at 6 months or Dose 3 at 12 months.

Hypothesis: The Geometric mean titers in the 12 month test group (T) are non-inferior to the usual timing control group (C):

H0: δ ≤ -δ0 versus H1: δ > -δ0 where δ = log (GMTT )- log (GMTC) and δ0 is the pre-specified non-inferiority margin

DETAILED DESCRIPTION:
1. Specific Aims and Overview: The investigators propose a randomized, open label trial of HPV vaccine among males 18-24 years old, comparing an on-time administration of the third dose with delayed administration of the third dose. All participants would receive the first and second doses according to schedule. They would be randomized to either Dose 3 at 6 months or Dose 3 at 12 months.

Blood would be drawn for titers at twice from all participants: pre-dose 1 and one month post Dose 3.

No cytology studies or DNA studies will be conducted.

1.1 Aims:

1. Determine if delay in the third dose is immunologically non-inferior to the standard administration schedule (1 month post-dose 3).
2. Determine the side effect profile of a delayed third dose, in comparison to the standard schedule.
3. Determine the preference and compliance of the men for the timing of the third dose.

1.2 Hypothesis for non- inferiority:

The GMTs in the test group (T) are non-inferior to the usual timing control group (C):

H0: δ ≤ -δ0 versus H1: δ > -δ0 where δ = log (GMTT )- log (GMTC) and δ0 is the pre-specified non-inferiority margin.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-26

Exclusion Criteria:

* Hospitalization within the past year
* Previous HPV vaccination

  >/=5 sexual partners (i.e., insertive intercourse) No other drug studies within 30 days of proposed HPV vaccination
* History of genital warts
* Immunosuppression
* Other vaccines within 8 days of proposed HPV vaccination
* Hypersensitivity to yeast or HPV vaccine components
* Known autoimmune disorders
* Receipt of immunoglobulins or blood product within 90 days of enrollment (may defer until 90 days completed)
* Serious Adverse Reaction to HPV vaccine

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Zimmerman, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Zimmerman RK, Nowalk MP, Lin CJ, Fox DE, Ko FS, Wettick E, Cost G, Hand L, Hayes J, Michaels M. Randomized trial of an alternate human papillomavirus vaccine administration schedule in college-aged women. J Womens Health (Larchmt). 2010 Aug;19(8):1441-7. doi: 10.1089/jwh.2009.1753. PMID 20629576
- [Result] Lin CJ, Zimmerman RK, Nowalk MP, Huang HH, Raviotta JM. Randomized controlled trial of two dosing schedules for human papillomavirus vaccination among college age males. Vaccine. 2014 Feb 3;32(6):693-9. doi: 10.1016/j.vaccine.2013.11.098. Epub 2013 Dec 14. PMID 24342252
- [Derived] Zimmerman RK, Lin CJ, Raviotta JM, Nowalk MP. Do vitamin D levels affect antibody titers produced in response to HPV vaccine? Hum Vaccin Immunother. 2015;11(10):2345-9. doi: 10.1080/21645515.2015.1062955. PMID 26176493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2010 through May 2011, college age men, ages 18-25 years, were recruited using a variety of strategies including fliers, class announcements, recommendations by university health centers, emails to campus organizations, bus and campus newspaper advertisements, and targeted Facebook® advertisements.
Pre-assignment Details: Exclusion criteria were: >4 lifetime sexual partners, health problems that would interfere with the immune response or ability to complete the study, a hospitalization during the past year, hypersensitivity to yeast or HPV vaccine components, inability to complete appointments, received HPV vaccine or immunosuppressive medications.
Groups:
- 12 Month Administration: Administration of 3rd dose at 12 months
  quadrivalent human papillomavirus vaccine : 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 12 months
- 6 Month Administration: 3rd dose administration at 6 months
  quadrivalent human papillomavirus vaccine : 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 6 months
Period: Overall Study
Arm/Group | 12 Month Administration | 6 Month Administration
Started | 111 | 109
Dose 2 | 110 | 108
Dose 3 | 101 | 107
Final Blood Draw | 97 | 107
Completed | 97 | 107
Not Completed | 14 | 2
Not completed — Lost to Follow-up | 14 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 Month Administration | 6 Month Administration | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 101 | 100 | 201
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (2.3) | 21.4 (2.2) | 21.3 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 109 | 220
Region of Enrollment [Number; unit: participants]
  United States | 111 | 109 | 220

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity After Dose 3
Description: Geometric mean titer (GMT) and 95% confidence intervals around titer 1 month after dose 3 in per protocol population, comparing the two groups.
Time Frame: 1 month after dose 3 (e.g., month 7 if third dose at 6months or month 13 if third dose at 12 months)
Population: Intention-to-treat
Measure: Geometric Mean (95% Confidence Interval); unit: mM units/ml
Arm/Group | 12 Month Administration | 6 Month Administration
Number analyzed (Participants) | 111 | 109
mM units/ml
  HPV 6 | 1063 [793 to 1312] | 794 [565 to 1009]
  HPV 11 | 1961 [1480 to 2403] | 1043 [689 to 1382]
  HPV 16 | 6186 [4947 to 7315] | 4555 [3243 to 5788]
  HPV 18 | 1049 [728 to 1350] | 709 [338 to 1103]
Statistical Analysis 1: Comparison: 12 Month Administration vs 6 Month Administration; The primary endpoint would demonstrate noninferiority if the upper bound of the 95% two-sided confidence interval (CI) of the ratio of GMT for Standard schedule group divided by that of Alternate schedule group is <1.5; Test type: Non-Inferiority or Equivalence — Sample size: (1 + 1/u)(Zα + Zβ)2 σ2 /[log (RGMT) -δ0] u= ratio of the size of the Standard schedule to Alternate schedule groups (u =1, for equal size groups); one-sided alpha (0.025)/4 for multiplicity of serotypes. Average log-transformed and geometric mean titers (GMTs) with a two-sided 95% confidence interval of the ratio of the GMTs were used. Non-inferiority is determined if upper bound GMT ratio of standard group to alternate group < 1.5; largest upper bound GMT ratio = 0.82 — Non-inferiority is determined if upper bound GMT ratio of standard 6 month group to alternate 12 month group < 1.5

2. Secondary Outcome: Compliance With 3rd Dose
Description: Determine the compliance of the men for the timing of the third dose.
Time Frame: at 3rd dose (i.e., at month 6 or month 12, depending on arm)
Measure: Number; unit: participants
Arm/Group | 12 Month Administration | 6 Month Administration
Number analyzed (Participants) | 111 | 109
participants | 97 | 107

3. Secondary Outcome: Safety Profile
Description: Total proportion of side effects reported after any dose, compared by arm.
Time Frame: 1 week after vaccination
Population: Intention-to-treat
Measure: Number; unit: percentage of doses with side effects
Groups:
- Group With Administration of 3rd Dose at 12 Months: Group with administration of 3rd dose at 12 months
  quadrivalent human papillomavirus vaccine : 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 12 months
- Group With Administration of 3rd Dose at 6 Months: Group with administration of 3rd dose at 6 months
  quadrivalent human papillomavirus vaccine : 0.5 mL of quadrivalent HPV vaccine at enrollment, 2 months, and 6 months
Arm/Group | Group With Administration of 3rd Dose at 12 Months | Group With Administration of 3rd Dose at 6 Months
Number analyzed (Participants) | 101 | 107
percentage of doses with side effects | 28.9 | 24.4
Statistical Analysis 1: Comparison: Group With Administration of 3rd Dose at 12 Months vs Group With Administration of 3rd Dose at 6 Months; null hypothsesis: no difference in proportion of side effects reported between groups; Test type: Superiority or Other; p = 0.26, Chi-squared

ADVERSE EVENTS:
Arm/Group | 12 Month Administration | 6 Month Administration
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/109
Other Adverse Events (participants affected / at risk) | 0/111 | 0/109

LIMITATIONS AND CAVEATS:
Drop-out rates higher in the Alternate group; however, sample size was met for all HPV types. The effect of the Alternate dosing schedule on long-term clinical outcomes is unknown. One syncopal episode related to phlebotomy prior to vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No